CLINICAL TRIAL: NCT04762654
Title: Turkish Version of the Faces Version of the Modified Child Dental Anxiety Scale: Evaluation of Validity and Reliability
Brief Title: Turkish Version of Modified Child Dental Anxiety Scale
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sema Aydınoglu, Associated professor, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 985
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Behavior; Child, Only; Anxiety, Dental
MeSH Terms: conditions — Behavior; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Modified Child Dental Anxiety Scale (MCDASf) — The MCDASf is self-reported dental anxiety measure effective among children aged 5-12 years.11 The scale has eight questions about 'going to the dentist generally,' 'having teeth examined,' 'teeth being scraped and polished,' 'injections in the gum,' 'fillings,' 'having a tooth taken out,' 'being put to sleep for treatment,' and 'having a mixture of gas and air that will help you feel comfortable for treatment but will not make you sleep.' The scores of each question ranged from 1 'relaxed' to 5 'very worried.' The scores are also represented by cartoon faces varied according to emotions and anxiety levels. The total scores can range from 8 to 40.

SUMMARY:
Background: The faces version of the Modified Child Dental Anxiety Scale (MCDASf) is less time consuming and an easy to understand tool for measuring dental anxiety. The aim of this study was to develop the Turkish version of MCDASf and to analyze its validity and reliability.

DETAILED DESCRIPTION:
The internal consistency reliability was determined by calculating Cronbach's alpha (n=300). Intraclass correlation coefficients (ICCs) were calculated for test-retest reliability (n=67). Construct validity was determined by comparing with the Venham Picture Test (VPT). The factor structure was examined using exploratory factor analysis (EFA). Confirmatory factor analysis (CFA) was used for the dimensionality. The cut-off points of the Turkish version of MCDASf were plotted using a receiver operating characteristic (ROC) curve.

ELIGIBILITY:
Inclusion Criteria:

* aged between 6-12 years, intellectual sufficiency to complete the questionnaire, and voluntariness to take part in the study. Also, only children whose parents were willing to participate were included

Exclusion Criteria:

* Children who had mental or physical disorders, cooperation problems or dental pain were excluded from the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children who presented for the first time to the Faculty of Dentistry in Rize
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
The Turkish version of MCDASf is a reliable scale that meets psychometric properties. | for six months from the beginning of the study
  The reliability of the Turkish version of MCDASf was assessed using the Cronbach alpha coefficient and Intraclass correlation coefficients (ICCs). Cronbach alpha coefficient scores vary from 0 to 1. Values higher than 0.70 are considered acceptable, and values higher than 0.80 are considered good internal consistency reliability. ICC values lower than 0.40 indicate poor agreement, 0.41-0.60 moderate agreement, 0.61-0.80 good agreement, and values higher than 0.80 show excellent agreement.
The Turkish version of MCDASf is a valid scale that meets psychometric properties. | for six months from the beginning of the study
  The validity of the Turkish version of MCDASf was assessed using The Venham Picture Test (VPT). The VPT includes eight cards that have two figures; one shows an anxious child, the other is not anxious. All cards are shown in order. For the selection of anxious and non-anxious figures, 1 and 0 points are recorded, respectively. The total scores can range from 1 to 8.

CONTACTS AND LOCATIONS:
Overall Officials: Ipek Arslan, Dr, Principal Investigator — Recep Tayyip Erdogan University Training and Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Recep Tayyip Erdogan University Training and Research Hospital, Rize
  - Sema Aydinoğlu, Rize

IPD SHARING:
Plan to Share IPD: Undecided